CLINICAL TRIAL: NCT02845180
Title: In-Vivo Assessment of Adipose Allograft Extracellular Matrix in Abdominoplasty Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Musculoskeletal Transplant Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: MTF 16-02-02
Record Dates: First submitted 2016-03-03; First posted 2016-07-27 (Estimated); Last update posted 2018-09-19 (Actual); Status verified 2016-07

CONDITIONS: Obesity
Keywords: lipectomy; panniculectomy
MeSH Terms: conditions — Obesity | interventions — Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 3 Mo. Post AAM Injection (Experimental): Injection. Adipose Allograft Extracellular Matrix (AAM). Panniculectomy post injection, 3 months.
  Interventions: Procedure: Adipose Allograft Extracellular Matrix (AAM) Injection
- 6 Month Post AAM Injection (Experimental): Injection. Adipose Allograft Extracellular Matrix (AAM). Panniculectomy post injection, 6 months.
  Interventions: Procedure: Adipose Allograft Extracellular Matrix (AAM) Injection

INTERVENTIONS:
Procedure: Adipose Allograft Extracellular Matrix (AAM) Injection — Injection followed by surgery

SUMMARY:
The purpose of this study is to assess local tissue reaction and retention of an adipose allograft extracellular matrix at 3 or 6 months post-injection into the subcutaneous abdominal tissue of healthy volunteers scheduled to undergo elective panniculectomy.

DETAILED DESCRIPTION:
This is a prospective, randomized, two arm, single center study to assess adipose tissue development and retention when an implantable allograft adipose matrix ('AAM') is injected in the abdominal subcutaneous tissue of healthy volunteers undergoing elective standard-of-care panniculectomy. This study will enroll ten (10) subjects. These subjects will be randomized to one of two study arms. Arm 1 will consist of five (5) subjects who will receive injections of AAM to be followed clinically for three (3) months duration, and arm 2 will consist of five (5) subjects who will receive injections of AAM to be followed clinically for six (6) months duration. At the point of completion of each arm, 3 or 6 months, the injected tissue will be surgically removed as part of the panniculectomy procedure. Samples of the AAM injected tissue areas and surrounding tissue will be obtained and processed for histologic evaluation.

ELIGIBILITY:
Inclusion Criteria

* Scheduled to undergo elective abdominoplasty.
* Able to provide informed consent.
* Able to understand and comply with the study design and are willing to return for all of the research required follow-up visits.
* BMI great than or equal to 23 and less than or equal to 35.
* Thickness of subcutaneous tissue on abdominal wall is at least 2cm thick.
* If a female, must test negative on a urine pregnancy test.
* If a female, must be willing to utilize an acceptable method of birth control (i.e., oral contraceptives, condom with spermicide, etc.) for the duration of the study.

Exclusion Criteria:

* Thickness of subcutaneous tissue on abdominal wall is less than 2cm thick.
* Previous liposuction at intended sites of treatment.
* Actively taking immunosuppressive therapy including systemic steroids (intranasal/inhaled steroids are acceptable).
* Actively receiving chemotherapy or radiation treatment.
* Subjects with a life expectancy of less than 9 months, terminal conditions or factors making follow-up difficult (e.g.; no fixed address, telephone, etc.)
* Subjects with intolerance to additional study-associated drugs/therapies (e.g.; lidocaine, etc.).
* Subjects with known coagulopathy.
* Subjects on chronic anticoagulants (e.g. Coumadin, etc.).
* Subjects who are pregnant, lactating or planning pregnancy during the study period.
* Subjects with abnormal blood chemistry or any abnormal laboratory finding considered clinically significant in that it would deem the subject inappropriate for surgical procedures, as determined by the Investigator (i.e., CBC with Differential, platelets, comprehensive metabolic panel to include electrolytes, bun/creatinine, liver function test and coagulation tests).
* Subjects who have, as determined by the investigator, a history or clinical manifestations of significant renal, hepatic, cardiovascular, metabolic, neurologic, psychiatric, or other condition that would preclude participation in the study (e.g.; Type I and II diabetic patients).
* Subjects with known alcohol or narcotic drug dependency that is deemed to impact compliance.
* Subjects with diagnosed autoimmune disorders known to affect wound healing, such as Systemic Lupus Erythematosis (SLE), psoriasis, infection and inflammation (seborrheic dermatitis).
* Subjects currently enrolled in another investigational study.

Study Population Description: Patients scheduled to undergo elective abdominoplasty Sampling Method: Invitation to volunteer

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2018-06-15 (Actual); Study Completion 2018-06-15 (Actual)

PRIMARY OUTCOMES:
Histopathology evaluation for number of mature adipocytes via haematoxylin and eosin staining. | 6 months
  Change from baseline to 6 months in abdominal tissue samples using H & E staining

SECONDARY OUTCOMES:
Safety of allograft adipose matrix (AAM) injections as determined by the incidence of adverse events. | 6 months
  Ongoing analysis of adverse events collected for the duration of a subject's participation and ongoing aggregate analysis of all subjects' adverse events. These endpoints will not be tested statistically unless unusual or unexpected results are obtained.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pittsburgh, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: Undecided
Decision to be made at study site appointment

REFERENCES:
- [Background] Flynn LE. The use of decellularized adipose tissue to provide an inductive microenvironment for the adipogenic differentiation of human adipose-derived stem cells. Biomaterials. 2010 Jun;31(17):4715-24. doi: 10.1016/j.biomaterials.2010.02.046. Epub 2010 Mar 20. PMID 20304481
- [Background] Brown BN, Freund JM, Han L, Rubin JP, Reing JE, Jeffries EM, Wolf MT, Tottey S, Barnes CA, Ratner BD, Badylak SF. Comparison of three methods for the derivation of a biologic scaffold composed of adipose tissue extracellular matrix. Tissue Eng Part C Methods. 2011 Apr;17(4):411-21. doi: 10.1089/ten.TEC.2010.0342. Epub 2011 Feb 5. PMID 21043998
- [Background] Wu I, Nahas Z, Kimmerling KA, Rosson GD, Elisseeff JH. An injectable adipose matrix for soft-tissue reconstruction. Plast Reconstr Surg. 2012 Jun;129(6):1247-1257. doi: 10.1097/PRS.0b013e31824ec3dc. PMID 22327888
- [Background] Omidi E, Fuetterer L, Reza Mousavi S, Armstrong RC, Flynn LE, Samani A. Characterization and assessment of hyperelastic and elastic properties of decellularized human adipose tissues. J Biomech. 2014 Nov 28;47(15):3657-63. doi: 10.1016/j.jbiomech.2014.09.035. Epub 2014 Oct 7. PMID 25446266